CLINICAL TRIAL: NCT03592394
Title: Immersive Virtual Reality for Chronic Neuropathic Pain After Spinal Cord Injury: A Feasibility Trial
Brief Title: Virtual Reality for Chronic Neuropathic Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kathleen Friel (Other)
Responsible Party: Sponsor-Investigator, Kathleen Friel, Lab Director, Clinical Laboratory for Early Brain Injury Recovery, Burke Medical Research Institute
Organization: Burke Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRC527
Record Dates: First submitted 2018-05-17; First posted 2018-07-19 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatic IVR (s-IVR) (Active Comparator): This group will use an Immersive Virtual Reality (Gear VR) device to focus on encouraging disassociation between pain and visualization and movement of the affected limbs. Subjects in this group will be exposed to an IVR environment that cycles them through a series of stretching and mobility exercises for the affected limbs bilaterally.
  Interventions: Device: Immersive Virtual Reality (Gear VR)
- Distractive IVR (d-IVR) (Active Comparator): This group will use an Immersive Virtual Reality (Gear VR) device to focus on distracting the subject from the pain. Subjects in this group will be exposed to a variety of engaging landscape IVR environments, without the ability to visualize their own body.
  Interventions: Device: Immersive Virtual Reality (Gear VR)

INTERVENTIONS:
Device: Immersive Virtual Reality (Gear VR) — Immersing the user in a total visual environment.

SUMMARY:
The investigators hypothesize that SCI patients using immersive IVR training will show improved reduction of neuropathic pain that will outlast the training sessions and transfers into daily life.

DETAILED DESCRIPTION:
Neuropathic pain (NP) affects 40 to 70% of people with SCI and is a very disabling clinical condition. The definitions of NP as well as its neurophysiology are widely discussed in the literature. Many treatment options have been offered, but provide limited effects, leaving people with SCI with a reduced quality of life.

Pain is a very complex experience that depends strongly on cognitive, emotional, and educational influences. Despite intensive investigations, the cause of neuropathic pain often remains unknown. A careful assessment of the pain including the use of tools to objectively measure pain will help with the diagnosis and the quantification of the damage. These tools include: 1) Laboratory testing that uses quantitative tests and measures objective responses in neurophysiology, sensory evoked potentials...etc.; 2) Quantitative sensory testing, that tests the perception of pain in response to external stimuli; 3) Bedside examination: physicians assessment on location, quality and intensity of pain; 4) Pain questionnaires, depending entirely on the subject's self-reported experience.

When spinal cord injury occurs, the spinal somatosensory circuit is thought to generate aberrant nociceptive impulses that the brain interprets as pain. Thalamic circuits may also serve as amplifiers of nociceptive signals. Sensory deafferentation after injury to the spinal cord produces extensive and long-lasting reorganization of the cortical and subcortical sensory maps. It has been suggested that pain and phantom limb sensations are the consequence of those cortical plasticity change. Therefore, strategies aimed at reversing or modulating the somatosensory neural reorganization may be valuable alternative approaches to neuropathic pain. Immersive virtual reality (IVR) is an emerging approach to the treatment of neuropathic pain conditions in SCI. Despite promising initial studies, IVR therapy has not yet been made widely available to individuals with SCI, because equipment is expensive and can be difficult for clinicians to use, especially those with limited experience with technology. However, with the development of 'plug and play', low-cost IVR devices such as the Oculus Rift, Gear VR and Google Cardboard, IVR no longer requires such specific technical knowledge. As a result, IVR is now a feasible and affordable treatment option for neuropathic pain.

The investigators believe that IVR neurorehabilitation exploits the idea of inducing activation in action observation, motor imagery, and processing systems, which in turn, should activate downstream cortical areas involved in movement and motor imagery. Also, perturbations of the somatosensory system associated with central pain can be reversed or modulated by employing motor imagery and related task execution combined with visual illusions. The investigators hypothesize that SCI patients using immersive IVR training will show improved reduction of neuropathic pain that will outlast the training sessions and transfers into daily life.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic neuropathic pain at or below SCI level for at least 6 months following trauma or disease of the spinal cord;
* A pain intensity of at least 4 out of 10 in the numerical rating scale (NRS) in the Neuropathic Pain Scale (NPS) test at both screening (baseline) and randomization (pre-evaluation);
* Stable pharmacological treatment for at least 2 weeks prior to the study and throughout the trial;
* Incomplete lesion (American Spinal Injury Association Impairment Scale, AIS B, C or D; B= motor complete, sensory incomplete; C= sensorimotor incomplete with an average strength of the muscles below the level of the lesion <3, D= sensorimotor incomplete with average muscle strength >3);
* Cervical level of lesion (C2 to T1) with presence of pain in the upper extremities

Exclusion Criteria:

* Presence of severe pain of other origin, such as musculoskeletal pain
* Psychiatric or other neurological disorders
* Head injuries causing cognitive or visual impairment
* Severe vertigo
* Presence of potential risk factors for brain stimulation (TMS): history of seizures, presence of surgically implanted foreign bodies such as a pacemaker, metal plate in the skull, and metal inside the skull;
* Medically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropathic Pain Scale | Baseline compared with immediately after intervention, and 1 month follow up
  It includes 11 items, assessing global pain intensity, unpleasantness, and one item which allows the patient to describe the temporal aspects of their pain and its qualities in their own words. The remaining 8 items assess specific NP qualities: "Sharp," "Hot," "Dull," "Cold," "Sensitive," "Itchy," "Deep," and "Surface." This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention.

SECONDARY OUTCOMES:
Upper Extremity Motor Score (UEMS) | Baseline, immediately after intervention, and 1 month follow up
  Clinical measure of motor strength
Modified Ashworth Scale | Baseline, immediately after intervention, and 1 month follow up
  Measure of spasticity scored from 1 (no increase in tone) to 4 (rigid limb)
Spinal Cord Independence Measure (SCIM III) | Baseline, immediately after intervention, and 1 month follow up
  Measures patient's ability to complete activities of daily living
Beck Depression Inventory | Baseline, immediately after intervention, and 1 month follow up
  Self-report measuring characteristic attitudes and symptoms of depression
Immersive Tendencies Questionnaire (ITQ) | Baseline, immediately after intervention, and 1 month follow up
  Measures an individual's sense of engagement and involvement in an activity
The Presence Questionnaire | Baseline, post-intervention, and 1 month follow up
  Measure of presence (ex: selective attention, involvement, immersive response, etc)
Patient's Global Impression of Change | Baseline, immediately after intervention, and 1 month follow up
  Evaluates both motor function and pain with no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7).
Transcranial Magnetic Stimulation | Baseline, immediately after intervention, and 1 month follow up
  Assess brain reorganization, output and responsiveness as determined by motor threshold, motor evoked potential and amplitude of response.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, PhD, Study Director — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.